CLINICAL TRIAL: NCT01339754
Title: Salvage Therapy With Trabectedin in Metastatic Pancreatic Adenocarcinoma: A Single-Arm Phase II Trial
Brief Title: Trabectedin in Treating Patients With Metastatic Pancreatic Cancer After First-Line Chemotherapy
Acronym: PACT-18
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000698981; PACT-18 (Other: IRCCS San Raffaele); 2010-024287-17 (EudraCT Number)
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trabectedin (Experimental): 1.3 mg/mq as a 3 hour continuous infusion every three weeks until progression
  Interventions: Drug: trabectedin

INTERVENTIONS:
Drug: trabectedin — 1.3 mg/mq as a 3 hour continuous infusion every three weeks
  Other Names: YONDELIS
Drug: trabectedin — 1.3 mg/mq as a 3 hour continuous infusion every three weeks until progression
  Other Names: ET 743

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as trabectedin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well trabectedin works in treating patients with metastatic pancreatic cancer after first-line chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the therapeutic activity of trabectedin, in terms of progression-free survival (PFS) rate at 6 months, in patients with metastatic pancreatic adenocarcinoma progressed after gemcitabine-containing first-line chemotherapy.

Secondary

* To assess the safety profile of this drug.
* To assess the response rate and response duration.
* To assess the overall survival of these patients.
* To assess the PFS rate at 9 and 18 weeks.
* To perform blood, plasma, and tumor tissue sampling for biological studies, in order to identify biomarkers predictive for resistance or sensitivity to trabectedin, and to characterize the impact of pharmacogenomic and pharmacokinetic profile on anti-tumor activity in translational research studies.

OUTLINE: Patients receive trabectedin IV over 3 hours on day 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Blood samples and tumor tissue are analyzed for identifying biological markers predictive for resistance to treatment and pharmacogenomic and pharmacokinetic profiling on anti-tumor activity in translational research studies.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas
* Metastatic disease progressed after 1 prior gemcitabine-contained chemotherapy

  * May be given with neoadjuvant, adjuvant, or palliative therapy
* Measurable disease according to RECIST criteria
* No symptomatic brain metastasis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Bone marrow, liver, and kidney function normal
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe comorbidities, including any of the following:

  * Cardiac disease
  * History of psychiatric disability
* No other prior or concurrent malignancy except surgically cured carcinoma in-situ of the cervix, basal cell or squamous cell carcinoma of the skin, and other neoplasms without evidence of disease for ≥ 5 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior second-line chemotherapy
* No other concurrent chemotherapy or target therapy
* No concurrent treatment with other experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 6 months | every 9 weeks
  CT scan

SECONDARY OUTCOMES:
Safety profile | every 3 weeks
  outpatient visit, laboratory findings
Response rate and response duration | every 2 months
  CT scan
Overall survival | every 3 weeks during therapy, every 2-3 months thereafter
  outpatient visit, phone interview
PFS rate at 9 and 18 weeks | every 9 weeks
  CT scan
Identify biomarkers predictive for resistance or sensitivity to trabectedin | at trial start
  tissue, blood, serum collection
Impact of pharmacogenomic and pharmacokinetic profile on anti-tumor activity | based on a pre-definid sample collection schedule
  blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy